CLINICAL TRIAL: NCT00880633
Title: EUS Staging Accuracy of Periampullary Neoplasms: a Retrospective Review
Brief Title: Endoscopic Ultrasound Staging of Periampullary Neoplasms: Retrospective
Status: Completed | Type: Observational
Sponsor: Indiana University (Other)
Responsible Party: Dr. Julia LeBlanc, Indiana University
Other Study IDs: 0703-58
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2011-02-17 (Estimated); Status verified 2011-02

CONDITIONS: Periampullary Neoplasms
Keywords: EUS; periampullary neoplasms

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this retrospective study is to determine the degree to which a biliary stent affects EUS staging accuracy of ampullary tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be identified retrospectively through an existing Indiana University Medical Center EUS database and pathology database.
* Patients with and without biliary stents will be included.

Exclusion Criteria:

* Patients that were suspected to have ampullary tumors but who were ultimately found to have a normal ampulla will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Retrospective review of patients who have already undergone an EUS at this institution.
Sampling Method: Non-Probability Sample
Dates: Start 2007-04; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
The presence of a biliary stent decreases EUS staging accuracy due to the intervening shadow artifacts

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Hospital, Indianapolis, Indiana, United States